CLINICAL TRIAL: NCT02024022
Title: A Comparison of Bowel Prep Quality and Patient Satisfaction in Outpatients Undergoing Colonoscopy Preparation With Either a Standard Bowel Preparation or an Individualized Approach Using Sodium Picosulphatge/Magnesium Citrate or 4L Polyethylene Glycol Preparation Regimens
Brief Title: A Multicenter Single-blind Comparison Between Standard and Individualized Approach in Bowel Preparation Before Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, dr. Theodor Alexandru Voiosu, MD, gastroenterology resident, Clinical Hospital Colentina
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: COL GASTRO 4
Record Dates: First submitted 2013-12-23; First posted 2013-12-31 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Bowel Cleansing Process; Colonoscopy
Keywords: colonoscopy; bowel cleansing; polyethylene glycol; sodium picosulphate / magnesium citrate
MeSH Terms: interventions — Polyethylene Glycols; picosulfate sodium; magnesium citrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard approach (Active Comparator): patients will be randomized to one of the 2 currently used bowel preparation regimens in our clinic:
  * 4L split polyethylene glycol solution
  * split magnesium citrate/sodium picosulphate preparation regimen
  Interventions: Drug: Standard approach
- Individualized approach (Experimental): patients will receive either the 4L split polyethylene glycol bowel prep regimen or the sodium picosulphate/magnesium citrate split prep regimen according to personal characteristics assessed using a self-administered questionnaire (including bowel habits, the preference for large-volume preparation and education level)
  Interventions: Drug: Individualized approach

INTERVENTIONS:
Drug: Standard approach — bowel cleansing with either 4L PEG or sodium picosulphate/magnesium citrate
  Arms: Standard approach
Drug: Individualized approach
  Other Names: 4 L polyethylene glycol or sodium picosulphate / magnesium citrate
  Arms: Individualized approach

SUMMARY:
This study aims to compare a standard approach to bowel preparation for colonoscopy (using sodium picosulphate/magnesium citrate or 4lPEG) to an individualized approach where patients are assigned a specific regimen of either sodium picosulphate/magnesium citrate or 4lPEG depending on patient-related factors. The study aims to compare patient-related outcomes such as comfort levels during bowel cleansing and physician-related outcomes such as bowel prep quality in the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* all patients > 18 years of age undergoing elective colonoscopy on an outpatient basis

Exclusion Criteria:

* refusal to sign informed consent
* pregnancy
* advance kidney, liver or heart disease
* suspicion of malignant / benign stenosis of the digestive tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
bowel cleansing | 24 hours
  bowel cleansing as assessed during colonoscopy using 2 assessment scales (Boston bowel prep scale, and a 1-4 semiquantitative scale)

SECONDARY OUTCOMES:
patient comfort level during bowel cleansing | 24 hours
  patient pain levels on a 0-10 visual analogue scale during the bowel cleansing process

CONTACTS AND LOCATIONS:
Overall Officials: Theodor Voiosu, MD, PhD, Principal Investigator — Clinical Hospital Colentina
Locations (3):
- Romania (3):
  - Colentina Clinical Hospital, Bucharest
  - Institutul Regional de Gastroenterologie si Hepatologie prof. dr. Octavin Fodor, Cluj-Napoca
  - Spitalul CFR, Cluj-Napoca

REFERENCES:
- [Background] Voiosu T, Ratiu I, Voiosu A, Iordache T, Schipor A, Baicus C, Sporea I, Voiosu R. Time for individualized colonoscopy bowel-prep regimens? A randomized controlled trial comparing sodium picosulphate and magnesium citrate versus 4-liter split-dose polyethylene glycol. J Gastrointestin Liver Dis. 2013 Jun;22(2):129-34. PMID 23799210